CLINICAL TRIAL: NCT03646162
Title: Randomized, Double-blind, Placebo Controlled, Dose Finding Phase 2 Study Comparing Oral Daily Dosing of VERU-944 to Ameliorate the Vasomotor Symptoms Resulting From ADT in Men With Advanced Prostate Cancer
Brief Title: Study of VERU-944 to Ameliorate Hot Flashes in Men With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V72203
Record Dates: First submitted 2018-08-17; First posted 2018-08-24 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — Zuclomiphene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Veru-944 10 mg (Experimental): Veru-944 10 mg daily
  Interventions: Drug: Veru-944
- Veru-944 50 mg (Experimental): Veru-944 50 mg daily
  Interventions: Drug: Veru-944
- Placebo (Placebo Comparator): Placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Veru-944 — Treat hot flashes (vasomotor symptoms) in men with advanced prostate cancer on ADT
  Other Names: Zuclomiphene citrate
  Arms: Veru-944 10 mg; Veru-944 50 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo controlled, dose finding Phase 2 study comparing oral daily dosing of VERU-944 after a week of loading (daily dosing) with placebo to ameliorate the vasomotor symptoms resulting from androgen deprivation therapy in men with advanced prostate cancer

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo controlled, dose finding study of VERU-944 to treat hot flashes (vasomotor symptoms) in men with advanced prostate cancer on ADT. The study will have four arms with 30 subjects per arm. The subjects participating in the study will have advanced prostate cancer and will be undergoing androgen deprivation therapy (ADT) with a luteinizing hormone releasing hormone (LHRH) therapy (agonist or antagonist) for at least the three months prior to randomization and be experiencing regular moderate to severe hot flashes while on ADT. Subjects will all continue to receive ADT and will be randomized to receive, for the first four days, a loading dose followed by daily doses of placebo or VERU-944 (10 mg, 50 mg or 100 mg) orally for a total period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Be over 18 years of age;
2. Be able to communicate effectively with the study personnel;
3. Have histologically confirmed prostate cancer;
4. Have been treated with an LHRH agonist or LHRH antagonist for at least the 3 months prior to randomization;
5. Be continued on an LHRH agonist or LHRH antagonist throughout this study;
6. Have experienced hot flashes for at least one month prior to study entry;
7. Have moderate or severe vasomotor symptoms (hot flashes) (defined as a minimum of 4 moderate to severe hot flashes per day or 12 per week at baseline);
8. ECOG performance status of 0 to 2
9. Be willing to uses electronic data capture for the relevant medical events

   • Must be at least 80% compliant during the screening period
10. Subjects must agree to use acceptable methods of contraception:

    * If their female partners are pregnant or lactating, acceptable methods of contraception from the time of the first administration of study medication until 6 months following administration of the last dose of study medication must be used. Acceptable methods are: Condom used with spermicidal foam/gel/film/cream/suppository. If the subject has undergone surgical sterilization (vasectomy with documentation of azospermia), a condom with spermicidal foam/gel/film/cream/suppository should be used.
    * If the male subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e., barrier method of contraception], surgical sterilization (vasectomy with documentation of azospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom used with spermicidal foam/gel/film/cream/suppository).
    * If the female partner has undergone documented tubal ligation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository) should also be used.
    * If the female partner has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used.
11. Subject is willing to comply with the requirements of the protocol through the end of the study.

Exclusion Criteria

1. Have a serum total testosterone concentration > 50 ng/dL at screening;
2. Known hypersensitivity or allergy to estrogen or estrogen like drugs;
3. Any disease or condition (medical or surgical) which might compromise the hematologic, cardiovascular, endocrine, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk;
4. Subjects with a personal history of abnormal blood clotting or thrombotic disease, including venous or arterial thrombotic events such as a history of stroke, deep vein thrombosis (DVT), and/or pulmonary embolus (PE);
5. Any subjects, as determined by a central laboratory, that have a:

   * Factor V Leiden gene mutation
   * Prothrombin gene mutation
6. Uncontrolled symptomatic congestive heart failure (NYHA Class III - IV), unstable angina pectoris, cardiac arrhythmia, or uncontrolled atrial fibrillation;
7. History of MI
8. The presence of consistently abnormal laboratory values which are considered clinically significant. In addition, any subject with liver enzymes (ALT or AST) above 2 times the upper limit of normal, total bilirubin above 2 times the upper limit of normal, or serum creatinine above 1.5 times the upper limit of normal will NOT be admitted to the study;
9. Received an investigational drug within a period of 90 days prior to enrollment in the study;
10. Received the study medication (VERU-944) previously;
11. Have previously taken within 6 months prior to screening or are currently taking diethylstilbestrol, other estrogens;
12. Currently taking gabapentin, estrogen, diethylstilbestrol, medroxyprogesterone acetate, clomiphene, selective serotonin reuptake inhibitors (SSRIs), other treatments for hot flashes
13. Recent hospitalization for more than 24 hours (within 30 days of screening);
14. Recent surgery (within 30 days of screening);
15. Have been previously diagnosed or treated for active cancer (other than prostate cancer or non-melanoma skin cancer) within the previous five years;
16. Have a BMI >40.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 93 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barnette, Study Chair — Veru Inc.
Locations (24):
- United States (24):
  - Gen1 Research, Glendale, Arizona
  - Tower Urology, Los Angeles, California
  - Urology of San Bernardino, San Bernardino, California
  - The Urology Center of Colorado, Denver, Colorado
  - Foothills Urology, Golden, Colorado
  - Universal Axon Clinical Research, Doral, Florida
  - Medical Research Center, Miami, Florida
  - North Idaho Urology, Coeur d'Alene, Idaho
  - First Urology, Jeffersonville, Indiana
  - Regional Urology LLC, Shreveport, Louisiana
  - Chesapeake Urology, Towson, Maryland
  - Coastal Urology, Brick, New Jersey
  - Premier Urology Group, Edison, New Jersey
  - Advance Urology, Elmont, New York
  - AccuMed Research, Garden City, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Medical Professionals, Syracuse, New York
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Urologic Consultants, Bala-Cynwyd, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Houston Urology Partners, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Urology of Virginia, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Started | 31 | 31 | 31
Completed | 26 | 27 | 30
Not Completed | 5 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 31 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 9 | 20
  >=65 years | 26 | 23 | 22 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (5.79) | 70.6 (8.84) | 69.1 (8.05) | 70.2 (7.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 30 | 30 | 31 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 9 | 10 | 31
  White | 18 | 20 | 21 | 59
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 31 | 91
Moderate to Severe Hot Flashes [Mean (Standard Deviation); unit: Percentage hot flashes moderate severe] | 41.5 (36.52) | 29.7 (22.2) | 33.7 (20.23) | 34.9 (26.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Moderate to Severe Hot Flashes at 6 Weeks
Description: Percentage of change in frequency of moderate to severe hot flashes at 6 weeks
Time Frame: 6 weeks
Population: Percentage of change in frequency of moderate to severe hot flashes at week 6
Measure: Mean (Standard Deviation); unit: Percentage of change in frequency
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Number analyzed (Participants) | 26 | 27 | 30
Percentage of change in frequency | -19.72 (8.840) | -42.24 (8.196) | -46.59 (7.760)

2. Secondary Outcome: Percentage Change in Severity of Moderate to Severe Hot Flashes at 6 Weeks
Description: Change in severity of moderate to severe hot flashes compared to baseline at 6 weeks
Time Frame: 6 weeks
Population: Percentage change in severity of moderate to severe hot flashes compared to baseline at 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Number analyzed (Participants) | 23 | 25 | 27
percentage of change | -0.21 (0.386) | -0.31 (0.416) | -0.35 (0.508)

3. Secondary Outcome: Change of Frequency of Moderate to Severe Hot Flashes at Week 12
Description: Mean change in frequency of moderate to severe hot flashes compared to baseline at weeks 12
Time Frame: Weeks 12
Population: Percentage of change from Baseline to Week 12
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Number analyzed (Participants) | 26 | 27 | 30
percentage of change | -39.94 (8.458) | -51.95 (8.574) | -52.70 (7.881)

4. Secondary Outcome: Change in Severity of Moderate to Severe Hot Flashes at Week 12
Description: Mean change in severity of moderate to severe hot flashes compared to baseline at week 12
Time Frame: Week 12
Population: Mean percentage change from baseline to week 12
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Number analyzed (Participants) | 26 | 27 | 30
percentage of change | -12.05 (5.014) | -16.93 (5.061) | -22.48 (4.674)

5. Secondary Outcome: Change in Bone Turnover Markers C-telopeptide (CTX)
Description: Change in C-telopeptide concentration at day 84 compared to baseline
Time Frame: 84 days
Population: Change in C-telopeptide concentration at day 84 compared to baseline
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Number analyzed (Participants) | 27 | 30 | 31
ng/L | 419.7 (262) | 362.1 (305.44) | 466 (347.3)

6. Secondary Outcome: Change in Bone Turnover Markers Alkaline Phosphatase
Description: Change in bone specific alkaline phosphatase at day 84 compared to baseline
Time Frame: 84 days
Population: Change in bone specific alkaline phosphatase at day 84 compared to baseline
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Number analyzed (Participants) | 28 | 30 | 31
ug/L | 13.89 (4.598) | 15.72 (22.468) | 13.12 (6.074)

7. Other Pre Specified Outcome: Change in Serum PSA
Description: Change in serum PSA concentration comparing baseline to day 30, baseline to day 60 and baseline to day 84 for each treatment group
Time Frame: 84 Days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Serum Total Testosterone
Description: Change in serum total testosterone concentration comparing baseline to day 30, baseline to day 60 and baseline to day 84 for each treatment group
Time Frame: 84 Days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Serum Free Testosterone
Description: Change in serum free testosterone concentration comparing baseline to day 84
Time Frame: 84 days
Population: Change in serum free testosterone concentration comparing baseline to day 84
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 29
ng/L | 1.16 (0.895) | 1.38 (4.873) | 1.0 (1.635)

10. Other Pre Specified Outcome: Change in Serum SHBG
Description: Change in serum SHBG concentration comparing baseline to day 30, baseline to day 60 and baseline to day 84 for each treatment group
Time Frame: 84 days
Population: Change in serum SHBG concentration comparing baseline to day 84
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
nmol/L | 55.7 (28.27) | 113.5 (60.53) | 54.1 (24.98)

11. Other Pre Specified Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)Sess Safety
Description: Incidence of Treatment-Emergent Adverse Events will be tabulated by MedDRA terms and system organ class. The incidence of AEs and the maximum intensity and frequency of AEs will be summarized. The intensity of AE will be graded according to CTCAE version 4. Changes from baseline will be computed and tested for significant change from baseline to day 114
Time Frame: 114 days
Reporting Status: Not Posted

12. Post Hoc Outcome: Post-hoc Analysis on the Percentage Change in Frequency of Moderate and Severe Hot Flashes From Baseline to Week 12; Exposure Response Assessment
Description: Post-hoc exploratory MMRM analysis was conducted to explore the effect of trough plasma concentration at Week12 on the change in frequency of moderate and severe hot flashes from Baseline to Week 12 in subjects with a BMI >25 kg/m2.
Time Frame: Day 84
Population: Subjects with a BMI >25 kg/m2 who had trough plasma concentrations ≥195 ng/mL vs <195 ng/mL Change in moderate and severe hot flash frequency at Week 12
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- PK ≥195ng/mL: Subjects who had trough plasma concentrations ≥195 ng/mL at Day 84 change in moderate and severe hot flash frequency at Week 12,
- PK <195 ng/mL: Subjects who had trough plasma concentrations <195 ng/mL at Day 84 change in moderate and severe hot flash frequency at Week 12,
Arm/Group | PK ≥195ng/mL | PK <195 ng/mL
Number analyzed (Participants) | 9 | 56
percentage of change | -77.60 (14.542) | -50.14 (5.842)

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Veru-944 10 mg | Veru-944 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30 | 2/31
Other Adverse Events (participants affected / at risk) | 7/30 | 16/30 | 11/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Veru-944 10 mg (N=30) | Veru-944 50 mg (N=30) | Placebo (N=31)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 — Atrial Fibrillation
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1 — Coronary Artery Disease
Appendicitis (Infections and infestations) | 0 | 1 | 0 — Appendicitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veru-944 10 mg (N=30) | Veru-944 50 mg (N=30) | Placebo (N=31)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — Constipation
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Dyspepsia
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — Flatulence
Nauseas (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Nauseas
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Abdominal Pain
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Abdominal Pain Upper
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Diarrhoea
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — gastroesophageal Reflux Disease
Urinary Tract Infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) — Urinary Tract Infection
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) — Nasopharyngitis
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Appendicitis
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Influenza
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Pneumonia
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Sinusitis
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Tooth Infection
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Upper Respiratory Tract Infection
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Arthralgia
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Muscle Spasms
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Arthritis
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Back Pain
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Myalgia
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Pain in extremity
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) — Headache
Balance Disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Balance Disorder
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Burning sensation
Disturbance in Attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Disturbance in Attention
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Dizziness
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Memory Impairment
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3) — Fatigue
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) — Oedema Peripheral
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — Pain
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) — Peripheral Swelling
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Hematuria
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Micturition urgency
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Nephrolithiasis
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Nocturia
Post micturition dribble (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Post micturition dribble
Renal Mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Renal Mass
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Anaemia
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Neutropenia
Atrial Fibrillation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Atrial Fibrillation
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Coronary artery disease
Vision Blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) — Vision Blurred
Cardiac Murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) — Cardiac Murmur
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) — Low density lipoprotein increased
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) — Hypertension
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Fall
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Insomnia
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Cough
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Alopecia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT03646162/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT03646162/SAP_001.pdf